CLINICAL TRIAL: NCT04539847
Title: Impact of Hearing Aid Technology on Self-reported Outcomes in Patients With Presbycusis - a Randomized Controlled Trial
Brief Title: Impact of Hearing Aid Technology on Self-reported Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: shoumoeller
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-06

CONDITIONS: Presbycusis, Bilateral
Keywords: hearing aid technology; presbycusis; self-reported outcome measures
MeSH Terms: conditions — Presbycusis

STUDY DESIGN:
Intervention Model Description: two-arm parallel assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-end hearing aid (Experimental): Patients will be fitted with premium level hearing aid technology
  Interventions: Device: High-end hearing aid
- Basic hearing aid (Experimental): Patients will be fitted with basic level hearing aid technology
  Interventions: Device: Basic hearing aid

INTERVENTIONS:
Device: High-end hearing aid — hearing aid with premium level of technology
  Other Names: Oticon; Resound; Widex
  Arms: High-end hearing aid
Device: Basic hearing aid — hearing aid with basic level of technology
  Other Names: Oticon; Resound; Widex
  Arms: Basic hearing aid

SUMMARY:
The study aims to investigate if the level of hearing aid (HA) technology has an impact on self-reported outcomes in patients with presbycusis in terms of overall IOI-HA scores, Factor 1, Factor 2 scores, SSQ scores, and the SSQ domains. The study explores if presbycusis patients report better outcomes with premium level HA technology compared to basic level HA technology. Further, the study investigates if premium level HAs provide more high-frequency gain than basic HAs using Real Ear Measurements.

DETAILED DESCRIPTION:
In hearing rehabilitation clinics today, the choice of hearing aid (HA) technology level is primarily based on the individual hearing care providers´ preferences. There is a lack of knowledge in which level of HA technology should be chosen for patients with presbycusis and if these patients will report higher benefit from more technologically advanced hearing aids. Therefore, this study aims to investigate if level of hearing aid technology has an impact on self-reported outcomes measures as the IOI-HA, SSQ, and 15-D questionnaire in patients with presbycusis.

The study was designed as a two-arm parallel randomized controlled trial. A subgroup of patients diagnosed with presbycusis and participating in the Danish National Better hEAring Rehabilitation (BEAR) project was invited to participate in the study.

Data was collected from the Department of Audiology at Odense University Hospital (OUH), Region of Southern Denmark.

All patients underwent a hearing examination which consisted of a pure-tone audiometry, bone-conduction thresholds at 250 Hz to 4 kHz, and a measure of word recognition scores (WRS) and speech reception thresholds (SRT) detecting the threshold at the 50% correct response level.

The questionnaires were sent to all patients two weeks prior to the first visit in clinic and included; a non-standardized health-related questionnaire containing questions on demographic details such as sex, age, HA experience, motivation and the SSQ questionnaire. The IOI-HA questionnaire was sent if patients were experienced HA users at the time of inclusion. All questionnaires were compiled and managed using Research Electronic Data Capture (REDCap) tools developed by Vanderbilt University, Nashville, Tennessee, United States (Harris et al. 2009, 2019) and is hosted by Odense Patient Explorative Network (OPEN) in the Region of Southern Denmark. Patients received the questionnaires through an online link generated by REDCap, but a paper-and-pencil version was also available if necessary when they entered the clinic.

Patients were randomized into two groups based on age, sex and WRS, and fitted with either a high-end or a basic level hearing aid.

Approximately two months after hearing aid fitting, a follow-up visit was scheduled where a Real Ear Measurement (REM) was carried out. The IOI-HA and SSQ questionnaires were re-sent to all patients two weeks prior the follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with presbycusis

Exclusion Criteria:

* Not being able to fill out questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
International Outcome Inventory for Hearing Aids | two months
  Hearing aid benefit questionnaire that consists of seven questions targeting different outcome domains.
  Each question is scored on a scale from 1 to 5 where a higher score indicates a better outcome.
Speech, Spatial, and Quality of hearing scale (the short form) | two months
  Hearing aid benefit questionnaire that consists of 12 questions targeting the hearing ability in different situations.
  Each question is ranked on a scale from 0 to 10 where a lower score indicates a greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper H Schmidt, PhD, MD, Principal Investigator — Odense University Hospital, Region of Southern Denmark

IPD SHARING:
Plan to Share IPD: No
All personal data will become anonymized and handled with full confidentiality in compliance with the Personal Data Processing Act and GDPR. The procedure of personal data processing will be reported to the Danish Data Protection Agency (Datatilsynet) in Odense University Hospital, Region of Southern Denmark.

REFERENCES:
- [Derived] Houmoller SS, Wolff A, Tsai LT, Narayanan SK, Hougaard DD, Gaihede ML, Neher T, Godballe C, Schmidt JH. Impact of hearing aid technology level at first-fit on self-reported outcomes in patients with presbycusis: a randomized controlled trial. Front Aging. 2023 Jun 1;4:1158272. doi: 10.3389/fragi.2023.1158272. eCollection 2023. PMID 37342862